CLINICAL TRIAL: NCT02978404
Title: A Phase II, Multi-centre Study, of Combining Radiosurgery and Nivolumab in the Treatment of Brain Metastases From Non-small Cell Lung Cancer and Renal Cell Cancer
Brief Title: Combining Radiosurgery and Nivolumab in the Treatment of Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16.206; OZM-080 (Other: CRO)
Record Dates: First submitted 2016-11-21; First posted 2016-12-01 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Clear-Cell Metastatic Renal Cell Carcinoma; Non Small Cell Lung Cancer Metastatic; Brain Metastases, Adult; Small Cell Lung Cancer; Melanoma
Keywords: radiosurgery; PD-1; Nivolumab
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Brain Neoplasms; Small Cell Lung Carcinoma; Melanoma | interventions — Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiosurgery and Nivolumab (Experimental): Interventions: Nivolumab (240mg IV q2week or 480mg IV q4week) and Radiosurgery (15-20 Gray (Gy) in 1 fraction)
  Upon entering this trial, patients with metastatic brain disease(s) will receive Nivolumab. One to 2 week after receiving the first dose of Nivolumab, radiosurgery will be delivered at doses ranging from 15 to 20 Gy in 1 fraction to the brain metastases to a maximum volume of 10 cubic centimeter.
  Interventions: Drug: Nivolumab; Radiation: Radiosurgery

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is administered to patients to a maximum of 2 year.
Radiation: Radiosurgery — Up to 10 cubic centimeter of brain metastases will be treated with radiosurgery. The dose of radiosurgery depends on the size of individual metastases.
  Other Names: SRS

SUMMARY:
Stereotactic radiosurgery (SRS) is increasingly administered as the sole treatment of brain metastases, in order to spare acute and long term side effects associated with whole brain radiotherapy. Local control of SRS treated lesions is good, but patients tend to develop additional brain metastases subsequently.

Nivolumab is a modulator of the immune system. Treatment with Nivolumab is associated with an increase in local control and survival in patients with non-small cell lung cancer and clear cell renal cell carcinoma. In the presence of Nivolumab, treatment of brain metastases with SRS may trigger an immune reaction against cancer. Therefore, the combination of SRS with Nivolumab may reduce the development of new brain metastases and improve patient survival.

The purpose of this study is to assess the effect of combining Nivolumab and SRS in controlling cancer progression. SRS will be administered to patients while they are receiving Nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ≥ 18 years of age
2. Willing and able to give written informed consent
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 within 28 days prior to registration
4. Radiation Therapy Oncology Group (RTOG) neurological function score of 0-1 within 28 days prior to registration
5. Histologic diagnosis of NSCLC, SCLC, Melanoma OR ccRCC
6. Stage IV cancer with brain metastases (Patients may have untreated primary disease)
7. Presenting with previously un-irradiated brain metastasis (10 cc maximum volume of brain disease based on the diagnostic screening MRI done within 28 days of registration))
8. Measurable/evaluable brain disease
9. Having received less than 4 lines of prior systemic treatments
10. Ability to be treated with either gamma knife or a linear accelerator based radiosurgery system
11. Ability to complete neurocognitive exams without assistance
12. Ability to complete QOL questionnaires with or without assistance
13. Screening laboratory values must meet the following criteria and should be obtained within 28 days prior to registration:

    * White Blood Cell (WBC) ≥ 2000/uL
    * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
    * Platelets≥ 100 x 109/L
    * Hemoglobin ≥ 90 g/L (may be transfused)
    * Serum creatinine ≤ 1.5 x Upper Limit of Normal (ULN) or Creatinine Clearance ≥ 50 ml/min (calculated -cockcroft-Gault)
    * Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤3 x ULN without liver metastasis,≤ 5 x ULN with liver metastases
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
14. Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (28 days plus the time required for Nivolumab to undergo five half-lives) after the last dose of investigational drug
15. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of Nivolumab
16. Women must not be breastfeeding
17. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving Nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of Nivolumab product. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception).

Exclusion Criteria:

1. Brain metastasis in the brainstem
2. Patients who experienced prior seizures are eligible, however patients should not have had a seizure within 7 days of registration without the use of corticosteroids.
3. All other cancer histology other than NSCLC or ccRCC
4. Patients who cannot undergo MRI
5. Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
6. Patients with a condition requiring systemic treatment with either corticosteroids including steroids used for treating peritumoral edema (> 50 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Drugs with a predisposition to hepatoxicity should be used with caution in patients treated with Nivolumab-containing regimen
8. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of Nivolumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
9. History of prior treatment with a CTLA-4, PD-1 or PD-L1 inhibitor, CD137 agonist, or anti-PD-L2.
10. Concomitant therapy with any of the following: IL-2, interferon, or other non-study immunotherapy regimens; immunosuppressive agents; other investigation therapies
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.
12. Known history of hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
13. History of allergy to study drug components.
14. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Intracranial progression-free survival | 1 year
  To evaluate whether the combination SRS with Nivolumab will improve the intracranial progression-free survival of patients.
  Response will be assessed as per RECIST version 1.1.

SECONDARY OUTCOMES:
Treated brain lesions control rate | 1 year
  Treated brain lesions control will be assessed as per RECIST version 1.1.
Overall survival after receiving Nivolumab. | 2 years
  Overall Survival is assessed at the end of the study at 2 years. A subject will be classified as either alive or dead due to any cause.
  The time to event will be calculated as the time from Day 1 until date of death.
  Day 1 is the date of 1st treatment consisting of an infusion of Nivolumab.
Maximum response rate of distant non-irradiated disease | 1 year
  Response will be assessed as per RECIST version 1.1.
Progression-free survival | 1 year
  Response will be assessed as per RECIST version 1.1.
Correlation between tumor PD-L1 expression and clinical outcomes | 1 year
  Tumor PD-L1 expression level will be correlated with patient overall response rate, loco-regional recurrence free survival and overall survival.
Patient quality of life | 1 year
  Quality of life will be assessed using the the Functional Assessment of Cancer Therapy - General (FACT-G) and the Brain Subscale (FACT-BR) questionnaires. A composite score will be obtained from the score of each subscale. Quality of life decline is the time to the first minimal important difference in the composite score from baseline.
Neurocognitive function, as measured by the HVLT-R | 1 Year
  Neurocognitive function will be assessed using the Hopkins Verbal Learning Test - Revised (HVLT-R). Neurocognitive failure is the time to the first failure on the assessments using the Reliable Change Index. Baseline neurocognitive function will be compared to the test results at 1 year using either a t-test or Wilcoxon-Mann-Whitney test, depending on the normality of the data.
Neurocognitive function, as measured by TMT | 1 year
  Neurocognitive function will be assessed using the Trail Making Test (TMT). Neurocognitive failure is the time to the first failure on the assessments using the Reliable Change Index. Baseline neurocognitive function will be compared to the test results at 1 year using either a t-test or Wilcoxon-Mann-Whitney test, depending on the normality of the data.
Neurocognitive function, as measured by COWA | 1 Year
  Neurocognitive function will be assessed using the Controlled Oral Word Association (COWA). Neurocognitive failure is the time to the first failure on the assessments using the Reliable Change Index. Baseline neurocognitive function will be compared to the test results at 1 year using either a t-test or Wilcoxon-Mann-Whitney test, depending on the normality of the data.
Acute and late toxicity of SRS + Nivolumab | 1 year
  Adverse events will be coded according to MedDRA. The results will be tabulated to examine their frequency, organ systems affected, severity, and relationship to study treatment.
  Terminology Criteria for Adverse Events (CTCAE) V4.03 will be used for grading of AEs. Investigators will provide their assessment of causality as 1) unrelated, 2) unlikely, 3) possibly related, 4) probably, or 5) definitely related.
Imaging indicators of response | 1 year
  Patient response to the treatment will be analysed using the Immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wong, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (4):
- Canada (4):
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec